CLINICAL TRIAL: NCT03941275
Title: SelectSecure 3830 Lead Imaging
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT18066
Record Dates: First submitted 2019-05-01; First posted 2019-05-07 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Heart Diseases
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subjects undergoing bi-plane fluoroscopy
  Interventions: Diagnostic Test: Bi-plane fluoroscopy

INTERVENTIONS:
Diagnostic Test: Bi-plane fluoroscopy — In vivo acquisition of biplane cine radiographic images of the market released Medtronic SelectSecure 3830 pacing lead

SUMMARY:
This study is designed to collect high-quality shoulder and intracardiac bi-plane fluoroscopic images during two standard arm motions on patients implanted with a market released SelectSecure 3830 lead for the purposes of developing a fracture reliability model.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at least 18 years of age
* Patient has a pacing, ICD or CRT system incorporating at least one SelectSecure 3830 lead in the right atrium or right ventricle
* Patients able and willing to attend imaging session
* Patients able and willing to give informed consent
* Pacing capture threshold and pacing impedance of the lead are within normal range at the time of enrollment
* Patient must be able to accomplish arm flexion and adduction past 90 degrees

Exclusion Criteria:

* Subjects who require a legally authorized representative to obtain consent
* Subjects with exclusion criteria required by local law (e.g. age, breastfeeding)
* Pregnant women, or women of child bearing potential and who are not on a reliable form of birth control
* Subjects that were implanted with a pacing, ICD, CRT device and/or cardiac leads less than three months ago

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects of both genders, 18 years of age and older that are currently implanted with at least one SelectSecure 3830 lead, regardless of device type and who meet all inclusion and no exclusion criteria are eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Collect high quality shoulder and intracardiac bi-plane fluoroscopic cine images of the SelectSecure 3830 pacing lead. | approximately 30 minutes
  Fluoroscopic cine images will be collected in conjunction with a specialized calibration object. When imaging data is processed and analyzed it will characterize the time-varying lead shape changes.

SECONDARY OUTCOMES:
Acquire accelerometer-based motion data | approximately 30 minutes
  During fluoroscopy of the two standard arm motions, accelerometer-based motion data will be collected which will allow matching of arm position with lead shape based on the fluoroscopic images.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Heart Center Research, Huntsville, Alabama
  - Iowa Heart Center, West Des Moines, Iowa
  - Associates in Cardiology PA, Silver Spring, Maryland
  - Lourdes Cardiology Services, Voorhees Township, New Jersey

IPD SHARING:
Plan to Share IPD: No